CLINICAL TRIAL: NCT00912678
Title: Prospective Randomized Controlled Trial to Compare a Calcineurin Inhibitor Free Immunosuppression With a Low Dose Tacrolimus Based Immunosuppression in "Old for Old" Kidney Transplantation.
Brief Title: Minimizing Immunosuppression in Old for Old Kidney Transplantation
Acronym: ESP-CNI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: Astellas Pharma GmbH (Industry)
Responsible Party: Prof. Dr. Lutz Fricke, MD PhD, University of Luebeck Medical School, Medical Clinic I, Transplant Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESP-2004-1
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation; Old for old kidney transplantation; European senior program; Calcineurin inhibitor free immunosuppression
MeSH Terms: interventions — Mycophenolic Acid; Steroids; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MMF and Steroid Group (Active Comparator): Group of Patients randomized to MMF and Steroid maintenance immunosuppression after 3 months (Tacrolimus withdrawal)
  Interventions: Drug: MMF (Cellcept) and Steroids
- Low-Dose Tacrolimus Group (Active Comparator): Patients randomized to withdrawal of MMF after 3 months and maintenance immunosuppression with low-dose tacrolimus and Steroids
  Interventions: Drug: Tacrolimus (Prograf)

INTERVENTIONS:
Drug: MMF (Cellcept) and Steroids — Prograf was withdrawn completely after randomization, MMF and steroids were given.
  Other Names: Prograf; CellCept
  Arms: MMF and Steroid Group
Drug: Tacrolimus (Prograf) — After randomization CellCept was withdrawn completely, low-dose tacrolimus was given.
  Other Names: Prograf
  Arms: Low-Dose Tacrolimus Group

SUMMARY:
Kidney transplantation in the elderly is a challenge since patient's co-morbidity and the decreased injury threshold of older grafts may limit the benefits of transplantation in these patients. To compare favourable effects between low dose tacrolimus (LD-Tac) and mycophenolate-mofetil (MMF) in this patient population the investigators conducted a one year prospective multicenter randomized controlled trial. 90 kidney transplant recipients > 65 years with cadaveric grafts (> 65 years) from 5 centers were enrolled and received baseline immunosuppression with daclizumab induction (1 mg/kg) at day one and day 14, LD-Tac (trough level 5-8 µg/ml), MMF (1-2 g/d) and steroids. After three months, patients were centrally randomized either to MMF (1-2 g/d) and steroids (23 patients) or to LD-Tac and steroids. Follow-up visits were performed every 4 weeks up to one year. Protocol biopsies were performed after one year. The investigators' primary hypothesis is that the biopsy proven rejection rate in the MMF group is not significantly different compared to the LD-Tac group after one year. The investigators' secondary hypothesis is that graft function in the MMF group (reflected by the glomerular filtration rate and protocol biopsy result) is superior to the graft function in the LD-Tac group.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a cadaveric kidney transplant (first or re-transplant)
* Patients must met the criteria of the EUROTRANSPLANT program
* Organ allocation with the framework of EUROPEAN SENIOR PROGRAM (ESP) by EUROTRANSPLANT
* Written consent

Exclusion Criteria:

* Not fulfilled inclusion criteria
* Cadaveric kidney from "non heart beating donors"
* One or more than one steroid resistant acute rejections within the first 3 weeks after transplantation
* Two or more than two steroid sensitive rejections (more than 2 administered steroid boli) within the first 3 weeks after transplantation
* Tacrolimus trough level > 10ng/ml in three consecutive measurements
* Allergy against macrolide antibiotics or tacrolimus
* Systemic steroid therapy at study entry not related to transplantation
* History of Malignancy
* Clinical relevant uncontrolled infections, heavy diarrhea, vomiting or active ulcer disease
* Patients who are enrolled in other clinical studies or were enrolled in other clinical studies 28 days before transplantation
* Patients under medication not approved by the German Ministry of Health

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2002-03; Primary Completion 2006-07 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Acute rejection rate | One year

SECONDARY OUTCOMES:
Graft function | One year

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Fricke, MD, PhD, Principal Investigator — University of Luebeck
Locations (5):
- Germany (5):
  - Transplant Center Cologne (Koeln-Mehrheim), Cologne, Cologne
  - University of Essen - Transplant Center, Essen, Hesse
  - Charite- Transplant Center - Campus Mitte, Berlin, State of Berlin
  - Charite - Transplant Center - Virchow Clinic, Berlin, State of Berlin
  - University of Luebeck, Transplant Center, Lübeck

REFERENCES:
- [Background] Vincenti F, Kirkman R, Light S, Bumgardner G, Pescovitz M, Halloran P, Neylan J, Wilkinson A, Ekberg H, Gaston R, Backman L, Burdick J. Interleukin-2-receptor blockade with daclizumab to prevent acute rejection in renal transplantation. Daclizumab Triple Therapy Study Group. N Engl J Med. 1998 Jan 15;338(3):161-5. doi: 10.1056/NEJM199801153380304. PMID 9428817
- [Background] Ducloux D, Motte G, Billerey C, Bresson-Vautrin C, Vautrin P, Rebibou JM, Saint-Hillier Y, Chalopin JM. Cyclosporin withdrawal with concomitant conversion from azathioprine to mycophenolate mofetil in renal transplant recipients with chronic allograft nephropathy: a 2-year follow-up. Transpl Int. 2002 Sep;15(8):387-92. doi: 10.1007/s00147-002-0403-3. Epub 2002 Aug 21. PMID 12221456
- [Background] Friemann S, Feuring E, Padberg W, Ernst W. Improvement of nephrotoxicity, hypertension, and lipid metabolism after conversion of kidney transplant recipients from cyclosporine to tacrolimus. Transplant Proc. 1998 Jun;30(4):1240-2. doi: 10.1016/s0041-1345(98)00226-7. No abstract available. PMID 9636504
- [Background] Pohanka E, Bechstein WO, Berlakovich G, Binet I, Friemann S, Heemann U, Kliem V, Sperschneider H, Stangl M, Ringe B. [Dosage and monitoring of tacrolimus after kidney transplantation]. Dtsch Med Wochenschr. 2000 May 12;125(19):608-11. No abstract available. German. PMID 11320722